CLINICAL TRIAL: NCT06333145
Title: The 90% Effective Dose (ED90) of Remimazolam Anesthesia Induction in Drug-induced Sleep Endoscope in Adult: an up and Down Sequential Trial
Brief Title: ED90 of Remimazolam Anesthesia Induction in Drug-induced Sleep Endoscopy in Adults
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDRA
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Effect of Drug
Keywords: Drug-induced Sleep Endoscopy; remimazolam; ED90
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal group (Experimental): BMI: ≥18.5 and <24
  Interventions: Drug: Remimazolam
- overweight group (Experimental): BMI: ≥24 and <30
  Interventions: Drug: Remimazolam
- obese group (Experimental): BMI: ≥30
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Exploring ED90 induced by remimazolam anesthesia in adults of different BMI groups undergoing drug-induced sleep endoscopy
  Other Names: Remimazolam besylate

SUMMARY:
Exploring the ED90 of remimazolam in Drug-induced Sleep Endoscopy in adults at different BMI groups.

DETAILED DESCRIPTION:
Exploring the ED90 of remimazolam in Drug-induced Sleep Endoscopy in adults at different BMI groups, to provide a more scientific medication scheme for sedation in Drug-induced Sleep Endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-65 years old, 2. ASA Ⅰ-Ⅲ level; 3. Sign an informed consent form.

Exclusion Criteria:

* 1.A history of central nervous system diseases, cognitive disorders, mental disorders, or communication disorders; 2.serious cardiovascular, respiratory, liver or kidney disease; 3.Anticipated need for tracheal intubation or laryngeal mask; 4.Allergic to benzodiazepines and opioids; 5.Those who have taken sedative, analgesic or antidepressant drugs within 24 hours; 6.Abnormal liver and kidney function; 7.Recently participated in other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ramsey Sedation Scale | 1 day
  Using the Ramsey Sedation Scale scoring table ranging from 1-6 to evaluate if the sedation is successful
  1point: Patients are anxious, restless or irritable; 2point: Patients cooperative, well-oriented and quiet; 3point: Patients fall asleep and respond only to commands; 4point: Patients fall asleep and respond quickly to eyebrow taps or loud auditory stimuli; 5point: Patients fall asleep and are blunt to respond to eyebrow taps or loud auditory stimuli; 6point: Patients fall asleep and do not respond to the above stimuli.

SECONDARY OUTCOMES:
Time records | 1 day
  Anesthesia time, induction time, surgical time, awakening time and recovery time
Use of drugs | 1 day
  The total amount of sedative and analgesic drugs used.
Respiratory suppression incidence | 1 day
  Respiratory frequency<8 times/min or SP02<90%
Incidence of Treatment-Emergent Adverse Events | 2 days
  Intraoperative blood pressure and heart rate changes: record the patient's intraoperative blood pressure, heart rate, and the use of related vasoactive drugs; Postoperative adverse reactions: such as hypertension, hypotension, tachycardia, gastrointestinal symptoms, postoperative restlessness, etc.
Incidence of PACU Adverse Reactions | 1 day
  Nausea and vomiting, pain (VAS score), hypotension, bradycardia, dizziness;

CONTACTS AND LOCATIONS:
Overall Officials: Aihua Du, Dr, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
You can request it from the main researcher.